CLINICAL TRIAL: NCT04304872
Title: Improving Physical Activity and Cardiac Rehabilitation Attendance Using Technology and Behavioral Economics
Acronym: IMPACT-CR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started due to delays with COVID and funding reallocation.
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 833631; 2P30AG034546-11 (NIH)
Record Dates: First submitted 2020-02-24; First posted 2020-03-11 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Cardiovascular Diseases
Keywords: cardiac rehabilitation; physical activity; wearable devices
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gamification Intervention (Experimental): Participants sign a pledge agreeing to try their best to meet their goals.
  Participants are entered into a game. Each week they receive 70 points. Each day, they are told their step count and points. If the step goal was met they keep their points, but if not, they lose 10 points. At the end of the week if they have at least 40 points they move up a level, but if not, they drop a level. Participants start in the middle of 5 levels.
  Participants choose a support partner who receives a weekly email with the participant's progress. The study group will hold a 3-way phone call with the participant and supportive sponsor to discuss ways they can help the participant meet their goal. At 6 weeks, the study group will have a follow up call if the participant is stuck in a lower level and restart them back at the middle level.
  Interventions: Behavioral: Gamification
- Loss-Framed Financial Incentive Intervention (Experimental): Participants are informed that each week that $14 is placed in a virtual account for them. Each day, the participant is informed of their step count on the prior day. If the step goal was achieved, the balance remains. Each day the goal is not achieved, the participant is informed that $2 was taken away.
  Interventions: Behavioral: Loss-Framed Financial Incentives
- Gamification and Loss-Framed Financial Incentive Intervention (Experimental): Participants receive both of the interventions described in the Gamification Intervention arm and the Financial Incentive Intervention arm.
  Interventions: Behavioral: Gamification; Behavioral: Loss-Framed Financial Incentives

INTERVENTIONS:
Behavioral: Gamification — Participants sign a pledge agreeing to try their best to meet their goals.
  Participants are entered into a game. Each week they receive 70 points. Each day they're told their step count and points. If the step goal was met they keep their points, but if not, they lose 10 points. At the end of the week if they have at least 40 points they move up a level, but if not, they drop a level. Participants start in the middle of 5 levels.
  Participants choose a support partner who gets a weekly email with the participant's progress. We hold a 3-way phone call with the participant and supportive sponsor to discuss ways they can help the participant meet their goal. At 6 weeks, we have a follow up call if the participant is stuck in a lower level and restart them back at the middle level.
  Arms: Gamification Intervention; Gamification and Loss-Framed Financial Incentive Intervention
Behavioral: Loss-Framed Financial Incentives — Participants are informed that each week $14 is placed in a virtual account for them. Each day the participant is informed of their step count on the prior day. If the step goal was achieved, the balance remains. Each day the goal is not achieved, the participant is informed that $2 was taken away.
  Arms: Gamification and Loss-Framed Financial Incentive Intervention; Loss-Framed Financial Incentive Intervention

SUMMARY:
The objective of this study is to test the feasibility of using behavioral economic interventions (gamification with and without loss-framed financial incentives) targeting daily steps counts to improve cardiac rehabilitation attendance.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of morbidity and mortality in the United States. Cardiac rehabilitation is a multifaceted physical activity program that incorporates medication adherence, smoking cessation, nutrition, and psychological counseling. Implementation of cardiac rehabilitation among those with cardiovascular disease (including ischemic heart disease, heart failure, and valvular heart disease) has been shown to increase physical activity and reduce cardiovascular mortality, morbidity, and hospital readmission rates. Cardiac rehabilitation carries a class I indication (standard of care) for post-acute coronary syndrome, post-percutaneous coronary intervention, in patients undergoing coronary artery bypass grafting/valve surgery, in patients with stable angina, and in patients with chronic heart failure per American College of Cardiology guidelines. Patient attendance and completion rates of a full regimen of cardiac rehabilitation therapy have been shown to be < 40% of those referred, depriving many eligible patients of the benefits of cardiac rehabilitation. The objective of this study is to test the feasibility of using behavioral economic interventions targeting daily step goals using wearable activity monitors to improve cardiac rehabilitation attendance among patients already referred for cardiac rehabilitation. We will compare three groups of 30 patients each as follows: 1) behaviorally designed gamification with social support; 2) loss-framed financial incentives; and 3) behaviorally designed gamification with social support AND loss-framed financial incentives.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18;
* Ability to consent;
* Patients with diagnosis of stable angina, chronic systolic heart failure, post- percutaneous coronary intervention, post-coronary artery bypass grafting surgery, post-acute myocardial infarction, and post-valvular repair who were discharged after an inpatient admission within the last 12 months;
* Smartphone or tablet compatible with application for the wearable activity tracking device;
* Independence Blue Cross health insurance coverage.

Exclusion Criteria:

* Conditions that would make participation infeasible such as inability to provide informed consent, illiteracy or inability to speak, read, and write English;
* Already enrolled in another study targeting physical activity;
* Medical condition preventing participation in a physical activity program;
* Prior or ongoing enrollment in cardiac rehabilitation;
* Baseline step count > 7,500 steps per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of cardiac rehabilitation sessions attended during intervention | Baseline to 12-week intervention period
  The primary outcome is the number of CR sessions attended during the 12-week intervention period.

SECONDARY OUTCOMES:
Proportion of patients that attend 30 of the 36 cardiac rehabilitation sessions during intervention | Baseline to 12-week intervention period
  The secondary outcome includes the proportion of patients that attend at least 30 of the 36 CR sessions during the 12-week intervention period.
Change in mean daily step counts from baseline to 12-week period | Baseline to 12-week intervention period
  The secondary outcomes include the change in daily step counts from baseline to the 12-week intervention period.

OTHER OUTCOMES:
Proportion of participants that identified a support partner | Baseline to 12-week intervention period
  We will explore measures of intervention acceptability and feasibility including the proportion of participants that identified a support partner.
Proportion of participants that completed the entire study | Baseline to 12-week intervention period
  We will explore measures of intervention acceptability and feasibility including the proportion of participants that completed the entire study.
Proportion of days that wearable device was used | Baseline to 12-week intervention period
  We will explore measures of intervention acceptability and feasibility including the proportion of days that the wearable device was used.

CONTACTS AND LOCATIONS:
Overall Officials: Neel Chokshi, MD, MBA, Principal Investigator — University of Pennsylvania
Locations (1):
- Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available.